CLINICAL TRIAL: NCT02501031
Title: Effect of Dietary Flaxseed on Circulating Sex Hormone Levels Among Post-menopausal Women - an Intervention Trial to Explore Flaxseed Intake as a Possible Breast Cancer Prevention Strategy
Brief Title: Flaxseed Intervention Study to Assess Sex Hormone Levels Among Post-Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Care Ontario (Other)
Collaborators: Canadian Breast Cancer Foundation, Ontario Region (funder) (Unknown); University of Toronto (Other); York University, Institute for Social Research (Unknown); Mount Sinai Services (Unknown); Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CBCF 2014-grant
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Flaxseed; Postmenopause; Hormones; Lignans; No Evidence of Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flaxseed (ground) (Experimental)
  Interventions: Dietary Supplement: Ground flaxseed
- Usual diet (No Intervention)

INTERVENTIONS:
Dietary Supplement: Ground flaxseed — 2 tablespoons of ground flaxseed taken daily for approximately 50 days.
  Arms: Flaxseed (ground)

SUMMARY:
The purpose of this study is to understand whether consuming flaxseed for approximately 50 days may beneficially affect the level of certain hormones in the blood thought to be involved in the development of breast cancer. This study will address the first steps toward the development of possible breast cancer prevention strategies. Differences in hormone levels (from blood samples) will be compared between two groups of women - those in the group assigned to eating ground flaxseed daily and those in the control group (with no change in diet).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate whether a dietary flaxseed intervention among post-menopausal women influences circulating levels of sex steroid hormones and estrogen metabolites (including estradiol, estrone, 2-hydroxy(OH)-/16-OH-estrone ratio, SHBG, testosterone, 2-MeOH-E1&-E2, 4-MeOH-E1&-E2) thought to be involved in the development of breast cancer.

SECONDARY OBJECTIVES:

II. Assess a) the effect of flaxseed intake on serum enterolignan levels (lignan biomarker), b) the relationship between serum enterolignan and sex hormone levels.

III. Describe adherence to the flaxseed intervention.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM 1: Participants take 2 tablespoons of ground flaxseed daily for approximately 50 days.

ARM 2: Participants maintain their usual diet for approximately 50 days.

All participants will complete a questionnaire and have their blood drawn at the beginning of the study (Day 0) and at the end of the study period (approximately Day 50).

ELIGIBILITY:
Inclusion Criteria:

1. Women residing in Toronto aged 57-64 years old, and post-menopausal.

Exclusion Criteria:

1. Consumers of flaxseed and soy (including supplements) in the past 6 months.
2. Consumers of sesame oil and sesame seeds in the past 6 months.
3. Women who took antibiotics orally in the past 6 months.
4. Women who took hormone replacement therapy or corticosteroids in the past month.
5. Non-English speaking.
6. Current chronic illnesses such as bowel disease (e.g. IBS - irritable bowel syndrome, or IBD - inflammatory bowel disease, such as Crohn's or ulcerative colitis), diabetes, heart disease (e.g. high cholesterol or high blood pressure and on medication for it), cancer, or another chronic illness.
7. Women who are currently taking blood thinners, such as Warfarin.

Ages: 57 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in circulating levels of sex steroid hormones at Day 0 (baseline) compared with ~Day 50 (end of study period) | Day 0 and ~Day 50

SECONDARY OUTCOMES:
Change in serum enterolignan levels at Day 0 (baseline) compared with ~Day 50 (end of study period) | Day 0 and ~Day 50

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cotterchio, PhD, Principal Investigator — Cancer Care Ontario and Dalla Lana School of Public Health, University of Toronto
Locations (1):
- Cancer Care Ontario, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No